CLINICAL TRIAL: NCT00641160
Title: A Phase 1 Study of the Safety, Pharmacokinetics, and Biological Activity of Metronomic Dosing With Orally Administered Vinorelbine Tablets in Subjects With Non-Hematologic Malignancies For Which There Are No Currently Accepted Therapies
Brief Title: Safety Study of Oral Vinorelbine in Subjects With Non-Hematologic Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Metronome Therapeutics (Industry)
Responsible Party: George Tidmarsh, MD, PhD, Metronome Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-CL002
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Nonhematologic Malignancies
Keywords: vinorelbine; metronomic dosing; oral administration; nonhematologic malignancies; pharmacokinetics
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental)
  Interventions: Drug: vinorelbine tartrate
- Cohort 2 (Experimental)
  Interventions: Drug: vinorelbine tartrate
- Cohort 3 (Experimental)
  Interventions: Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: vinorelbine tartrate — Dose Level #1 PO for at least 7 days
  Arms: Cohort 1
Drug: vinorelbine tartrate — Dose Level #2 PO for at least 7 days
  Arms: Cohort 2
Drug: vinorelbine tartrate — Dose Level #3 PO for at least 7 days
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to determine the safety of oral administration of vinorelbine once daily for at least 7 days. The study will be conducted in subjects with a non-hematologic malignancy for which there are no currently accepted therapies.

ELIGIBILITY:
Inclusion Criteria:

* capable of understanding study requirements and able to provide Informed Consent
* diagnosed with a non-hematologic malignancy for which there are no currently accepted therapies
* life expectancy at least 3 months
* agreement to use medically acceptable contraception throughout the study
* willing and able to comply with the protocol requirements

Exclusion Criteria:

* currently receiving systemic treatment for malignancy
* not yet recovered from the toxicity of prior therapies
* platelet count < 100,000 cells/mm3 within 7 days prior to study entry
* ANC < 1500 cells/mm3 within 7 days prior to study entry
* hemoglobin < 8.5 g/dL within 7 days prior to study entry
* AST and/or ALT > 2.5 X ULN within 7 days prior to study entry
* total bilirubin > 1.5 X ULN within 7 days prior to study entry
* creatinine clearance < 60 mL/min (Cockroft-Gault formula) within 7 days prior to study entry
* receipt of any investigational therapy within 3 weeks prior to study entry
* known history of HIV, HBV, and/or HCV infection
* clinically relevant active infection or serious co-morbid medical condition at study entry
* major surgery within 4 weeks prior to study entry
* other malignancy within 3 year prior to study entry
* pregnant or breast-feeding
* presence of a concomitant disease or condition which, in the opinion of the Investigator, could interfere with the conduct of the study or could put the subject at unacceptable risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by adverse events, physical examinations, clinical laboratory assessments, and vital signs | Assessed at each subject visit to the study center

SECONDARY OUTCOMES:
Pharmacokinetics of orally administered vinorelbine | Samples collected on Study Days 1, 2, and 8
Exploratory analysis of blood markers of biological activity | Blood samples collected at selected subject visits to the study center

CONTACTS AND LOCATIONS:
Overall Officials: George Tidmarsh, MD, PhD, Study Director — Metronome Therapeutics
Locations (1):
- Texas Oncology PA; Sammons Cancer Center, Dallas, Texas, United States